CLINICAL TRIAL: NCT05819268
Title: A Multi-site Feasibility Clinical Trial of Retraining and Control Therapy (ReACT), a Mind and Body Treatment for Pediatric Functional Seizures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Yale University (Other); Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Aaron Fobian, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-300010786
Record Dates: First submitted 2023-03-24; First posted 2023-04-19 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Functional Seizures; Convulsion, Non-Epileptic
MeSH Terms: conditions — Psychogenic Nonepileptic Seizures; Seizures

STUDY DESIGN:
Intervention Model Description: Children with FS will be enrolled and randomized to either ReACT or CATCH-IT therapies
Who Masked: Investigator
Masking Description: The PI, statistician and data manger will be blinded to treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ReACT Intervention (Experimental): During the initial visit participant will be randomized to either Retraining and Control Therapy (ReACT) or Competent Adulthood Transition with Cognitive Behavioral, Humanistic, and Interpersonal Training (CATCH-IT) intervention.
  ReACT includes 12 sessions with a therapist that will discuss a plan for managing FS.
  Participants will have 12 therapy sessions. The first session will be in-person which will last 2 hours and the subsequent 11 sessions will be conducted via video telehealth and each session will last 1 hour.
  Interventions: Behavioral: ReACT
- CATCH-IT Intervention (Active Comparator): During the initial visit participant will be randomized to either Retraining and Control Therapy (ReACT) or Competent Adulthood Transition with Cognitive Behavioral, Humanistic, and Interpersonal Training (CATCH-IT) intervention.
  CATCH-IT involves the parent and child completing CBT modules on the web-based CATCH-IT platform, and they will meet with a CATCH-IT coach 12 times to discuss the modules and plan how to apply this to their life and their FS.
  Participants will have 12 therapy sessions. The first session will be in-person which will last 2 hours and the subsequent 11 sessions will be conducted via video telehealth and each session will last 1 hour.
  Interventions: Behavioral: CATCH-IT

INTERVENTIONS:
Behavioral: ReACT — ReACT includes 12 sessions with a therapist that will discuss a plan for managing FS.
  Other Names: Retraining and Control Therapy
  Arms: ReACT Intervention
Behavioral: CATCH-IT — CATCH-IT involves the parent and child completing CBT modules on the web-based CATCH-IT platform, and they will meet with a CATCH-IT coach 12 times to discuss the modules and plan how to apply this to their life and their FS.
  Other Names: Competent Adulthood Transition with Cognitive Behavioral, Humanistic, and Interpersonal Training
  Arms: CATCH-IT Intervention

SUMMARY:
The purpose of this study is to assess the feasibility of conducting a future fully powered multi-site efficacy Randomized Controlled Trial (RCT) comparing two treatments for pediatric functional seizures (FS). In this study, 11-18-year-olds diagnosed with FS will be randomized to 12 sessions of Retraining and Control Therapy (ReACT) or Competent Adulthood Transition with Cognitive Behavioral, Humanistic, and Interpersonal Training (CATCH-IT) at 3 sites: University of Alabama at Birmingham, Yale School of Medicine/Yale New Haven Children's Hospital and Baylor College of Medicine/Texas Children's Hospital.

Feasibility of recruitment will be measured by the percentage of planned participant enrollment target obtained at each site and overall during the 18 months of planned enrollment. Acceptability will be assessed using the Acceptability Questionnaire. Participant retention will be measured by the percent of enrolled participants that complete the 2-month follow-up visit at each site and overall. For treatment fidelity assessment, 20% of each therapist's sessions will be randomly chosen and assessed for fidelity. Patient adherence will be measured in two ways: 1) the percent of ReACT or CATCH-IT sessions completed at each site and overall and 2) for ReACT, the percent of times participants report using the treatment plan during FS episodes (measured by FS diary) and for CATCH-IT, the number of times parents and children spend using CATCH-IT each week (measured by the CATCH-IT platform). These data will be used to support a future fully-powered multi-site RCT assessing the efficacy of ReACT for pediatric FS.

DETAILED DESCRIPTION:
This study aims to conduct a multi-site pilot feasibility Randomized Controlled Trial (RCT) at the University of Alabama at Birmingham, Yale College of Medicine/Yale New Haven Children's Hospital and Baylor College of Medicine/Texas Children's Hospital.

Participants with functional seizures (FS) will be screened for eligibility over a phone call and eligible participants will be invited for a baseline visit. Participants with FS and their parent/guardian will then complete a baseline visit and 2 follow-up visits via HIPAA-compliant Zoom, 1 in-person initial therapy session and 11 video telehealth follow-up therapy sessions via HIPAA-compliant Zoom.

During the initial baseline visit, participants and their family member/caregiver will complete several questionnaires assessing demographics, mood, relationships with friends and family, as well as past and current FS symptoms. Participants will receive a functional seizure diary to record all episodes during the course of the study. This visit will last about an hour and a half to 2 hours. They will then be randomized to 12 sessions of either Competent Adulthood Transition with Cognitive Behavioral, Humanistic, and Interpersonal Training (CATCH-IT) or Retraining and Control Therapy (ReACT). CATCH-IT involves the parent and child completing Cognitive Behavioral Therapy (CBT) modules on the web-based CATCH-IT platform, and they will meet with a CATCH-IT coach 12 times to discuss the modules and plan how to apply this to their life and their FS. ReACT includes 12 sessions with a therapist that will discuss a plan for managing FS. The first session for each intervention will be in-person with the subsequent 11 sessions conducted via video telehealth. Individual study teams from the 3 participating sites will conduct the ReACT or CATCH-IT interventions at their respective sites. The first therapy session will last about 2 hours and the subsequent 11 telehealth sessions will last about an hour.

There will be 2 follow-up visits via HIPAA-compliant Zoom which will follow the same protocol as the baseline visit. The first follow-up visit will be one week after the 12th therapy session, and the second follow-up visit will be two months after the 12th therapy session. Both these sessions will last about an hour.

Participants will also have the opportunity to undergo the therapy to which they were not randomized to after completing the 2-month follow-up after 12th therapy session.

There will be two long term follow-up visits via HIPAA-compliant Zoom, at 6 months after the final intervention session and at 12 months after the final intervention session where participants and parents will complete few questionnaires. Both these visits will last about 45 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ages 11-18
* Diagnosis of functional seizures
* Internet access for telehealth sessions and CATCH-IT

Exclusion Criteria:

* Comorbid epilepsy
* Less than 4 functional seizures per month
* Other paroxysmal nonepileptic events (e.g. hypoxic-ischemic phenomena, sleep disorders or migraine-associated disorders)
* Participation in other therapy
* Severe intellectual disability
* Severe mental illness (active delusions/hallucinations)

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Recruitment | 18 months
  Feasibility of recruitment will be measured by the percentage of the planned participant enrollment target obtained at each site and overall during the 18 months of planned enrollment. This includes any participant who completes informed consent/assent.
Acceptability | 18 months
  Acceptability will be assessed using the Acceptability Questionnaire. The Acceptability Questionnaire is based on a published theoretical framework for assessment of acceptability of healthcare interventions and assesses acceptability of being randomized to ReACT vs. CATCH-IT, acceptability of the treatment received and presence of treatment side effects associated with ReACT or CATCH-IT, including all side effects associated with mindfulness. For each reported side effect, the duration, tolerability, perceived unpleasantness, impact on functioning and acceptability based on treatment benefit will be obtained.
Participant Retention | 18 months
  With the goal of analyzing data from the subsequent efficacy trial with an intention-to-treat analysis, participant retention will be measured by the percent of enrolled participants that complete the 2-month follow-up visit at each site and overall.

SECONDARY OUTCOMES:
Participant Adherence | 18 months
  Patient adherence will be measured in two ways: 1) the percent of ReACT or CATCH-IT sessions completed at each site and overall and 2) for ReACT, the percent of times participants report using the treatment plan during FS episodes (measured by FS diary) and for CATCH-IT, the number of times parents and children spend using CATCH-IT each week (measured by the CATCH-IT platform).
Treatment Fidelity | 18 months
  Fidelity will be stratified by site and therapist/coach, such that 20% of each therapist/coach's sessions will be randomly chosen for fidelity assessment. The ReACT Fidelity Rating Scale includes assessment of the therapists' correct use of the ReACT Treatment Determination Tool, therapeutic alliance and empathy with the patient and family, development of opposing responses and use of motivators to reinforce progress. Fidelity to CATCH-IT sessions will be measured by the CATCH-IT coach fidelity scale, which assesses conduct of the motivational interview, review of the CATCH-IT sessions, therapeutic alliance and empathy with the patient and family.
Functional seizure frequency | 15 to 17 months
  FS Diaries will be completed in REDCap by parents and children to prospectively track FS frequency from 7 days prior to treatment through 12 months post treatment, including date, time, location, duration and nature of symptoms. Those in ReACT will report if they used their treatment plan for each FS and track each FS they prevented with the plan. They will retrospectively report FS for the 3 weeks prior to initial screening. Discrepancies in parent and adolescent report will be discussed and rectified to improve accuracy
Sense of Agency scale | 5 to 7 months
  Sense of Control Scale is a single question which asks, "How much control do you believe you have over your FS?" at baseline and post follow-up visits. Scores range from 0-3 with a higher score indicating no control over functional seizures.
Treatment Preference Questionnaire | Baseline Visit
  Treatment Preference Questionnaire will be completed before randomization to assess to which treatment the participant and parent prefer to be randomized. This is a single question which asks the participant "Which treatment would they prefer to be randomized to?".
Quality of Life in Epilepsy for Adolescents (QOLIE-AD-48) | 5 to 7 months
  Quality of Life in Epilepsy for Adolescents (QOLIE-AD-48) is a survey of health-related quality of life for children with epilepsy with higher scores indicating a poor quality of life. It is used in patients with FS by instructing them to consider their FS when asked about "seizures". Scores range from 0-100. This will be completed at baseline and at first 2 follow-up visits.
Revised Helping Alliance Questionnaire- II | 5 to 7 months
  Revised Helping Alliance Questionnaire-II is a 19-item scale will assess the therapist, children and parents' perception of the therapeutic alliance at at first 2 follow-ups. Scores ranges from 19-114 with a higher score indicating better therapeutic alliance.
The Credibility/Expectancy Questionnaire | 15 to 17 months
  The Credibility/Expectancy Questionnaire will be used to compare treatment expectancy between conditions. It measures how much the patient believes the therapy they are receiving will help to reduce their FS. This will be completed by parent and participant initially after being randomized, after the first session, fourth session, eighth session and at the follow-up visits.
Children's Somatic Symptoms Inventory (CSSI-24) | 15 to 17 months
  General somatic symptom complaints, higher scores indicate greater somatic complaints. Scores range from 0-140. Completed by participant and parent. Assessed at baseline visit and all 4 follow-up visits
Anxiety Sensitivity Index (ASI) | 15 to 17 months
  Assesses catastrophic symptom expectations; higher scores indicate greater anxiety. Completed by the parent. Assessed at baseline visit and all 4 follow-up visits
LEVEL 2-Somatic Symptom report adapted from the Participant Health Questionnaire | 5 to 7 months
  Measures symptom severity in children; higher scores indicate greater symptom severity. Completed by participant and parent. Assessed at baseline visit and at first 2 follow-up visits.
Functional Disability Inventory (FDI) | 5 to 7 months
  Completed by child and parent to measure physical functioning and disability in children with chronic pain; score ranges from 0-60, higher scores indicate greater perceived functional disability. Completed by participant and parent. Assessed at baseline visit and at first 2 follow-up visits
The Impact on Family Scale | 15 to 17 months
  Assesses parental perceptions of the impact of a child's medical condition on the family; higher scores indicate greater financial burden on the family. Assessed at baseline visit and all 4 follow-up visits.
The Revised Children's Anxiety and Depression Scale (RCADS) | 15 to 17 months
  Measures anxiety and depression symptoms in children; higher scores indicate increased symptom severity. Completed by participant and parent. Assessed at baseline visit and all 4 follow-up visits
Childhood Anxiety Sensitivity Index (CASI) | 15 to 17 months
  Assesses catastrophic symptom expectations; higher scores indicate greater anxiety. Score ranges from 18-54. Completed by participant. Assessed at baseline visit and all 4 follow-up visits
Healthcare Related Stigma Questionnaire | At Baseline visit
  Measures stigma in patients and their parents related to their interaction with health care providers; higher scores indicate greater stigma. Completed by participant and parent. Assessed at baseline visit.
Dysfunctional Attitude Scale (DAS-9) | 5 to 7 months
  Participant will complete this 9-item self-report measure that aims to determine stable negative attitudes that people with depression hold about themselves, the world, and their future. Assessed at baseline visit and at first 2 follow-up visits.
Behavior Rating Inventory of Executive Functioning (BRIEF) | 5 to 7 months
  Assesses executive function and self-regulation in children and teens. Completed by participant at baseline visit and at first 2 follow-up visits.
Beaver's Self-Report Family Inventory | 5 to 7 months
  This is a 36 item scale which assesses a family member's view of overall family competence. Completed by participant and parent. Assessed at baseline visit and at first 2 follow-up visits.
FND Locus of Control: Multidimensional Health Locus of Control (MHLC) Scales | 15 to 17 months
  Measures an individual's belief in his/her ability to control health outcomes. Form C of MHLC scale will be completed by participant at baseline and all 4 follow-up visits. Form A of MHLC scale will be completed by parent at baseline visit and first 2 follow-up visits.
Rosenberg Self-esteem scale | 5 to 7 months
  This is a 10-item scale measuring self esteem. Score ranges from 0-30 with low scores indicating low self-esteem. Completed by participant at baseline visit and at first 2 follow-up visits.
Mishel Uncertainty in Illness Questionnaire-Community Form (MUIS-C) | 5 to 7 months
  Participant will complete this 23-item scale which measures uncertainty about their diagnosis. Assessed at baseline visit and at first 2 follow-up visits.
Illness Cognitions Scale | 5 to 7 months
  Participant will complete this 17-item scale measuring the degree to which they align with the sick role. Assessed at baseline visit and at first 2 follow-up visits.
Center for Epidemiological Studies Depression Scale (CES-D) | 5 to 7 months
  Parent will complete this 10-item self-report depression inventory. Score ranges from 0 to 30 with higher scores indicating increasing levels of depression. Assessed at baseline visit and at first 2 follow-up visits.
Center for Epidemiological Studies Depression Scale for Children (CES-DC) | 5 to 7 months
  Participant will complete this 20-item self-report depression inventory. Score ranges from 0 to 60 with higher scores indicating increasing levels of depression. Assessed at baseline visit and at first 2 follow-up visits.
Parenting Style and Dimensions Questionnaire (PSDQ Short Version) | 5 months
  This is a 32-item scale assessing parenting style for self and partner. Completed by parent at baseline visit and 7-day follow-up visit.
Session Summary Sheet (SSS) | 5 to 7 months
  Assesses parent and participant's therapeutic relationship, mastery of skill and involvement in therapy session. Completed by therapist at each intervention visit.
FND Knowledge Questionnaire | 5 to 7 months
  Assesses parent and child's knowledge on FND. Completed by parent and child at baseline and at first 2 follow-up visits.
Other FND Symptoms Questionnaire | 15 to 17 months
  Assesses the intensity and frequency of FND symptoms other than FS. Completed by both child and parent at baseline and all 4 follow-up visits.
Clinical Global Impression | 5 months
  Assesses the patient's improvement in FS/FND which is due to treatment intervention. Completed by therapist during the 12 therapy sessions.
The Columbia Suicide Severity Rating Scale (C-SSRS) | 5 to 7 months
  Addresses the full range of suicidal thoughts and behaviors that suggest a person is at heightened risk of committing suicide. This includes previous suicide attempts, history of suicidal ideation and intent and last-minute aborted attempts due to a change of heart. Participants will complete the measure at baseline and at 7 days post and 2 months post follow-up visits
Single Quality of Life Question | 15 to 17 months
  Single quality of life question asks "Please rate your/your child's overall quality of life (i.e. your overall social, physical and mental wellbeing)". Completed by parent and participant at baseline and all 4 follow-up visits.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No